CLINICAL TRIAL: NCT03666533
Title: Transcranial Direct Current Stimulation for Post-stroke Gait Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N2620-R; 15036-H19 (Other Grant/Funding Number: Louis Stokes Cleveland VA Medical Center IRB)
Record Dates: First submitted 2018-09-04; First posted 2018-09-11 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Gait Impairment
Keywords: Gait therapy; transcranial Direct Current Stimulation (tDCS); Neuroplasticity; walking ability; brain stimulation; virtual reality
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: transcranial Direct Current Stimulation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS (Active Comparator): active tDCS plus gait training
  Interventions: Other: Active transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator): sham tDCS plus gait training
  Interventions: Other: Sham transcranial Direct Current Stimulation

INTERVENTIONS:
Other: Active transcranial Direct Current Stimulation — Active tDCS is combined with gait therapy. Gait therapy includes gait task practice in Virtual Reality setting and overground gait therapy
  Other Names: tDCS
  Arms: Active tDCS
Other: Sham transcranial Direct Current Stimulation — Sham tDCS is combined with gait therapy. Gait therapy includes gait task practice in Virtual Reality setting and overground gait therapy
  Other Names: Sham tDCS
  Arms: Sham tDCS

SUMMARY:
Stroke affects upwards of 800,000 Americans every year and has an enormous impact on the well-being of the American Veteran population with 6,000 new stroke admissions every year. Many of these stroke survivors are living with walking disabilities. Gait problems result in inability to function independently, high risk of falls and poor quality of life. Unfortunately, current gait rehabilitation treatments are limited and many stroke survivors do not achieve full recovery. Therefore, it is critical to develop new approaches to enhance gait rehabilitation methods. The investigators propose to evaluate a brain stimulation treatment called transcranial Direct Current Stimulation (tDCS) that can be added to physical therapy. tDCS has been applied for arm rehabilitation after stroke with positive results, but gait-related investigations are lacking. The investigators will test whether simultaneous tDCS and gait training produces greater improvement in walking abilities than gait training alone. Adjunct tDCS therapy may improve outcomes, and reduce cost of both rehabilitation and post-stroke care.

DETAILED DESCRIPTION:
Current rehabilitation methods fail to restore normal gait for many stroke survivors leading to dependence on others, recurrent falls, limitations in community ambulation and poor quality of life. The main objective of this study is to test both efficacy and neurophysiological mechanisms of a novel approach to treat persistent gait deficits after stroke with a combination of simultaneous non-invasive brain stimulation with transcranial Direct Current Stimulation (tDCS) and gait training. The investigators will enroll chronic stroke subjects (>6 months) with gait deficits. Subjects will be randomized to 10 sessions of either active tDCS+gait training or sham tDCS+gait training. Gait training will be accomplished in the treadmill-based Virtual Reality environment targeting longer single limb stance with the paretic limb. The primary outcome measure will be both gait speed and single limb stance duration. Other outcome measures will assess various components of gait-related functional domains. The study will also characterize neuroplastic brain changes in response to bihemispheric tDCS combined with gait training based on corticospinal excitability using motor evoked potentials and functional connectivity using resting state functional Magnetic Resonance Imaging (rs-fMRI).

ELIGIBILITY:
Inclusion Criteria:

* Medically and psychologically stable and at least 6 months after first ever unilateral stroke
* Cognition sufficiently intact to give valid informed consent to participate
* FMLE score >15; and ability to actively dorsiflex the paretic ankle in synergy (FMLE item II Flexor synergy-ankle dorsiflexion score 1).
* Sufficient endurance to participate in the study

Exclusion Criteria:

* Activity tolerance is insufficient to complete treadmill training
* Inability to produce a trace contraction of ankle dorsiflexors in synergy
* Normal ankle dorsiflexion/knee flexion on FMLE standing items (FMLE item IV score=4)
* Stroke affecting both sides
* Contraindications for rTMS according to the most recent TMS-use guidelines
* Contraindications for MRI
* Inability to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Pundik, MD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Pundik S, Skelly MM, McCabe JP, Salameh AI, Anderson T, Duncan KR, Hisel T, Carr SJA. Resting-State Functional Connectivity of Sensorimotor and Default Mode Networks and Lower Limb Performance in Chronic Stroke: A Cross-Sectional Study. Brain Behav. 2025 May;15(5):e70519. doi: 10.1002/brb3.70519. PMID 40329808

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 21 | 23
Completed | 19 | 21
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.7) | 67.7 (8.3) | 65.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 13 | 19 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 23 | 44
years post stroke, mean (SD) [Mean (Standard Deviation); unit: years] | 4.5 (3.4) | 4.5 (4.9) | 4.5 (4.2)
stroke type, Ischemic, n (count of participants) [Number; unit: participants] | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Gait Speed From Baseline (Meters/Second)
Description: Gait speed will be calculated based on Ten Meter Walk Test
Time Frame: baseline to post treatment (after 5 weeks of treatment)
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 19 | 21
meters/second | 0.16 (0.183) | 0.12 (0.141)

2. Secondary Outcome: Change From Baseline to Post Treatment on Timed up and go (Seconds)
Description: Gait function measure where individuals rise from a chair, walk 3 meters, turn around and return to sitting in the chair
Time Frame: baseline to post treatment (after 5 weeks of treatment)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 19 | 21
seconds | -6.93 (16.957) | -5.7 (8.314)

3. Secondary Outcome: Change From Baseline to Post Treatment in Functional Gait Assessment (Points)
Description: Functional gait measure where individuals walk under different conditions and are scored on a a 4 point scale for performance. 0-30 points; Higher score indicates better outcome
Time Frame: baseline to post treatment (after 5 weeks of treatment)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 19 | 21
points | 2.79 (3.047) | 2.38 (1.717)

4. Secondary Outcome: Change From Baseline to Post Treatment on Fugl Meyer Lower Limb
Description: Motor control measure for lower limb after stroke, items rated on a scale of 0-2. A higher score indicates better outcome. score range is 0-34 points.
Time Frame: baseline to post treatment (after 5 weeks of treatment)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 19 | 21
points | 2.26 (1.996) | 2.62 (2.334)

5. Secondary Outcome: Change From Baseline to Post Treatment on Gait Assessment and Intervention Tool
Description: Measure of gait coordination after stroke; lower score indicates better coordination; 0-62 points, with lower score indicating better outcome
Time Frame: baseline to post treatment (after 5 weeks of treatment)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 19 | 21
points | -2.42 (2.219) | -2.86 (2.78)

6. Secondary Outcome: Change in Asymmetry of Tibialis Anterior Muscle Motor Evoked Potentials From Baseline
Description: Motor Evoked Potential (MEP) is a measure of corticospinal excitability using Transcranial Magnetic Stimulation. We collected maximum MEP from the paretic and non-paretic limbs. Asymmetry of paretic and non-paretic MEPs was calculated as follows: non-paretic minus paretic divided by a sum of paretic and non-paretic. It is expected that therapy reduces asymmetry caused by stroke. We report number of participants with reduced asymmetry of paretic and non-paretic tibialis anterior muscle Motor Evoked Potential.
Time Frame: baseline to after 5 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 19 | 21
Participants | 9 | 8

ADVERSE EVENTS:
Time Frame: adverse event information for each participant was collected during their study participation (baseline to 6 week follow-up)
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 0/21 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT03666533/Prot_SAP_000.pdf